CLINICAL TRIAL: NCT02604654
Title: Phase IV Clinical Trial of Yiqitongluo Granule in the Treatment of Stroke With Qi-deficiency and Blood-stasis Syndrome
Brief Title: Effectiveness and Safety of Yiqitongluo Granule for Stroke
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yi Yang (Other)
Collaborators: Shineway Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor-Investigator, Yi Yang, Associated Dean of First Hospital of Jilin University, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SWYY-YQTLKL
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Last update posted 2021-08-25 (Actual); Status verified 2020-07

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yiqitongluo group (Experimental): Yiqitongluo granule 12g each time, 3 times a daily for 4 weeks.
  Interventions: Drug: Yiqitongluo granule

INTERVENTIONS:
Drug: Yiqitongluo granule — administered after dissolved

SUMMARY:
The purpose of the prospective study is to evaluate the effectiveness and safety of Yiqitongluo granule in the treatment of stroke with qi-deficiency and blood-stasis in more than sixy hospitals all over China.

ELIGIBILITY:
Inclusion Criteria:

* mild and moderate ischemic stroke patient with 4-25 NIHSS score
* stable patients within 1 week to 3 months
* sign informed consent before study

Exclusion Criteria:

* CT shows cerebral hemorrhage disease: such as hemorrhagic stroke, epidural hematoma, intracranial hematoma, ventricular hemorrhage, and subarachnoid hemorrhage
* severe disturbance of consciousness
* dysphagia
* TIA
* hemorrhagic diathesis
* patient with malignant tumor whose expected lifetime is less than 3 months
* allergic constitution
* gestation period, lactation period, woman with the possibility or plan of pregnancy
* those who participated in other clinical trials within 3 months or taking part in other clinical trials

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2197 (Actual)
Dates: Start 2015-12-29 (Actual); Primary Completion 2017-11-05 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Safety of Yiqitongluo for stroke measured by laboratory index | change from baseline laboratory index at 28(±7) days

SECONDARY OUTCOMES:
Effect of Yiqitongluo for stroke with mRS | 90(±7) days
  mRS: modified Rankin Scale
Effect of Yiqitongluo for stroke with syndrome of traditional Chinese medicine | 28(±7) days
Effect of Yiqitongluo for stroke with NIHSS | 28(±7) days
  NIHSS: the NIH stroke scale
Effect of Yiqitongluo for stroke with BI | 28(±7) days
  BI: Barthel Index
Effect of Yiqitongluo for stroke with EQ-5D | 28(±7) days
  The EQ-5D-3L essentially consists of 2 pages - the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, Study Chair — The First Hospital of Jilin University; Zhenni Guo, Study Director — The First Hospital of Jilin University